CLINICAL TRIAL: NCT01654432
Title: A Randomized Controlled Comparative Study of Ultrasound-guided Paravertebral Blocks as Part of a Multimodal Regimen for Ambulatory Breast Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Women's College Hospital (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-0004-B
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Breast Diseases
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- General anaesthesia and sham nerve block (Placebo Comparator): Breast cancer surgery under general anaesthesia
- Paravertebral Blocks (PVB) (Active Comparator): Breast cancer surgery under ultrasound-guided paravertebral blocks plus general anesthesia
  Interventions: Other: Paravertebral Blocks (PVB)

INTERVENTIONS:
Other: Paravertebral Blocks (PVB)
  Arms: Paravertebral Blocks (PVB)

SUMMARY:
General anesthesia and morphine based pain medicine analgesia has been the mainstay of practice in breast cancer surgery at Women's College Hospital. There is evidence to suggest that patients have a better recovery, with less pain and nausea and vomiting when nerve blocks or freezing of nerves are given in addition to a general anesthetic. Specifically for breast cancer surgery, evidence has suggested that the use of paravertebral blocks provide patients with a better quality of recovery after surgery. The aim of this study is to examine whether patients who receive the nerve blocks using an ultrasound machine in addition to general anesthesia have a better quality of recovery than patients who receive a general anesthetic alone. The hypothesis is that patients receiving ultrasound-guided paravertebral blocks (PVB) with propofol-based general anesthesia (GA) will have a better quality of recovery than patients receiving general anesthesia-opioid-analgesia. Quality of recovery will be assessed using a modification of the QoR-27, a validated instrument to assess postoperative recovery in an ambulatory surgical population.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer at stage T1-3, N0-2, M0, presenting for unilateral complete or partial mastectomy with or without sentinel lymph node dissection, with or without implant insertion
* ASA physical status I-II
* 18-85 years of age, inclusive
* BMI ≤ 35

Exclusion Criteria:

* Contraindications to paravertebral nerve block (e.g., allergy to local anesthetics, coagulopathy, malignancy or infection in the back area)
* Pregnancy
* History of alcohol or drug dependency/abuse
* History of significant psychiatric conditions that may affect patient assessment

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the quality of recovery at discharge as assessed by the QoR27 | Within 24 hours postoperatively
  The patient will be met with by the study coordinator, just before discharge to administer the Quality of Recovery Questionnaire (QoR27)
The primary outcome measure is the quality of recovery post operatively, as assessed by the QoR27 | on average between 24-48 hours postoperatively
  The patient will be contacted by the study coordinator, 2 days following their surgery to administer the Quality of Recovery Questionnaire (QoR27)
The primary outcome measure is the quality of recovery at discharge as assessed by the QoR27 | On average 72-96 hours post operatively
  The patient will be contacted by the study coordinator, 4 days following their surgery to administer the Quality of Recovery Questionnaire (QoR27)
The primary outcome measure is the quality of recovery post operatively as assessed by the QoR27 | On average 7-8 days postoperatively
  The patient will be contacted by the study coordinator, 7 days following their surgery to administer the Quality of Recovery Questionnaire (QoR27)

SECONDARY OUTCOMES:
Neuropathic pain | 6 months
  DN4

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Morgan, MD, CCFP, FRCPC, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada